CLINICAL TRIAL: NCT07217158
Title: Role of ROS and cAMP-PKA Signaling-related Biomarkers on Renal Disease Severity and Progression in ADPKD
Brief Title: Role of ROS and cAMP-PKA Biomarkers in ADPKD
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Maria V. Irazabal Mira, Principal Investigator, Mayo Clinic
Other Study IDs: 23-000116
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal Dominant Polycystic Kidney Disease (ADPKD); Oxidative stress; Antioxidant response; Mitochondria injury
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective is to determine the prognostic value of markers of ROS and cAMP-PKA signaling to assess disease severity and progression in patients with ADPKD.

DETAILED DESCRIPTION:
Individuals with ADPKD are born with normal renal function that is preserved for several decades. By the time the GFR starts to decline, most of the kidneys have been replaced by cysts. The median age of end-stage renal disease (ESRD) is 54 years for PKD1 and 74 years for PKD2, but the rate of disease progression varies widely among individuals. This variability, along with the maintenance of normal GFR until the late stages, represents a significant challenge for nephrologists in following these patients. It is difficult to predict disease progression or evaluate a new therapy based solely on renal function markers at an early stage. On the other hand, if new therapies are implemented when GFR starts to decline and most irreversible damage has occurred, they are less likely to be effective. Hence, identifying robust, early disease biomarkers predictive of GFR decline and disease progression is crucial.

The improvement of imaging techniques over the years has provided insights into the natural history of the disease and facilitated the observation of its structural progression. The Consortium for Radiologic Imaging Studies of PKD (CRISP) study has shown that in patients with ADPKD, the increase in kidney and cyst volumes directly correlates with GFR decline, underscoring the potential of TKV to monitor disease progression and as a primary or secondary endpoint in clinical trials for ADPKD. However, TKV has limitations as a biomarker, as it is fairly crude and does not fully capture the pathophysiological processes underlying the development and progression of the disease. Therefore, biomarkers related to the underlying molecular mechanisms may detect renal injury before permanent anatomical damage occurs.

The investigators' broad objective is to determine the value of NOX4, as well as surrogate markers for ROS, mitochondrial injury, and metabolic pathways, to assess disease severity and progression from early stages.

Participants in this study will have blood and urine samples collected to determine biomarkers of oxidative stress, antioxidant response, related metabolite levels, as well as kidney injury markers. In addition, an abdominal MRI will be performed to determine the patient's total kidney volume (TKV).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 15 - 70 years of age
* Previous diagnosis of ADPKD (based on Ravine et al. criteria)
* Class 1 A-E according to imaging classification
* estimated GFR> 45 mL/min/1.73 m2 (CKD-EPI)
* Ability to provide written, informed consent

Exclusion Criteria:

* Class 2, according to imaging classification
* A concomitant systemic disease affecting the kidney
* Diabetes mellitus
* Predicted urine protein excretion in >1 g/24 hrs. and or abnormal urinalysis
* Use of antioxidants, i.e., vitamins, Nrf2 activators
* Patients who are part of an interventional study or taking tolvaptan

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients with a previous diagnosis of ADPKD that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in height adjusted Total kidney volume (htTKV) | Baseline to 24 months
  TKV determined by MRI
Change in eGFR | Baseline to 24 months
  eGFR estimated by CKD-EPI
Baseline concentration of: NOX4, biochemical markers related to ROS, mitochondrial injury and metabolites as predictors of change in TKV and eGFR | Baseline to 24 months
  Biochemical markers determined by ELISA and/or biochemical assays, PCR, TKV determined by MRI, eGFR estimated by CKD-EPI.

SECONDARY OUTCOMES:
Change in concentration of: NOX4, biochemical markers related to ROS, mitochondrial injury and metabolites | Baseline to 24 months
  Biochemical markers determined by ELISA and/or biochemical assays, PCR,

CONTACTS AND LOCATIONS:
Overall Officials: Maria V. Irazabal, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No